CLINICAL TRIAL: NCT06423092
Title: Short-term Effectiveness of Music Therapy Songwriting on Mental Health Outcomes of At-risk Parents in the Neonatal Intensive Care Unit: an International Multicenter Mixed-methods Study.
Brief Title: Music Therapy Songwriting and Mental Health in Neonatel Intensive Care Unit (NICU) Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Aristizábal (Other)
Collaborators: Sanitas University (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Director, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 166-23 UNV
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mental Health Impairment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy songwriting + standard care (Experimental): The music therapy songwriting is a method frequently employed in music therapy sessions. This method involves the collaborative creation of lyrics and/or music with the participants. The intervention will consist of nine sessions, each of which will last approximately 30 to 45 minutes. Three sessions will be conducted per week until a minimum of six and a maximum of nine sessions are achieved.
  Interventions: Other: Music therapy songwriting
- Standard care (No Intervention): Standard care is the usual care provided to parents of newborns hospitalized in a neonatal intensive care unit (NICU). This care includes providing information about the baby's health status and recommendations during contact with the baby. Additionally, when a health professional identifies symptoms of mental health disturbance in the parents, they are referred to a mental health professional for appropriate management.

INTERVENTIONS:
Other: Music therapy songwriting — Session 1: The goal of the first music therapy session is to know the parents musically and to provide information about song creation. This is achieved by exploring their favorite songs. Options for creating a song (original song or song parody) are presented and possibilities for creating lyrics are discussed.
  Sessions 2-7: The structure of the song will be created and discussed with the parents. Parents will also be invited to include written messages from other family members in the lyrics if they wish. In each session, the developing welcome song is sung together with the parents, accompanied by the music therapist, who provides vocal or instrumental support.
  The final sessions (Sessions 8-9) are dedicated to singing the final version of the song with the parents and their infant. Should the parents desire, a final recording of the song will also be made and the digital songbook will be created.
  Arms: Music therapy songwriting + standard care

SUMMARY:
The mental health of parents of preterm newborns (PTNB) is negatively affected by prolonged hospitalization of the PTNB in the intensive care unit. This produces changes in the role of the parents and the bond with the newborn, leading to states of depression, anxiety, and stress. Several strategies, including music therapy, have been implemented to mitigate the negative impact on the parents' mental health.

The main objectives of the proposed trial are to determine whether Music Therapy (MT) songwriting combined with standard care (SC) during NICU stay is superior to SC alone in reducing the risk of postpartum depression in at-risk parents of preterm children at the end of treatment, and understand the lived experiences of participating parents who received music therapy for their mental health.

DETAILED DESCRIPTION:
This study employs a multicenter, mixed-method approach, with a quantitative component that will be a pragmatic parallel controlled randomized clinical trial (RCT) and a qualitative component that will include phenomenological study. The quantitative component will assess depression and anxiety, which will be evaluated with the Edinburgh Postnatal Depression Scale (EPDS) and the Generalized Anxiety Disorder Scale (GAD-7), respectively. Secondary outcomes will be resilience, coping, stress, and mental well-being. These outcomes will be measured in the first week of hospitalization (baseline measure) and then in weeks 1, 2, and 3 of the intervention. Changes in scores will be assessed to identify the effect, and mediating variables will be determined by multivariate analysis. Semi-structured interviews will be conducted on the parents' experience of music therapy songwriting for the baby.

The study will provide data on the effect of music therapy songwriting on the mental health of parents of neonates with brain injuries (PTNB) versus standard care and will document the lived experience of music therapy songs. The results may inform the standardization of this strategy in neonatal intensive care units (NICUs) to support and accompany parents and decrease the impact on their mental health.

ELIGIBILITY:
Inclusion Criteria:

* The study population consisted of parents/caregivers of newborns hospitalized in neonatal intensive care units (NICUs) with gestational ages of ≤32 weeks and expected hospitalizations of at least three weeks. In the case of a twin pregnancy, the firstborn infant was randomly assigned to one of the intervention groups, while both infants received the same treatment according to the outcome of randomization.
* Mother a total score of ≥10 and/or father a total score of ≥7 on the EPDS (Edinburgh Postnatal Depression Scale)
* Mother and/or father a total score of ≥8 on the GAD-7 (Generalized Anxiety Disorder Scale)

Exclusion Criteria:

* Parents/caregivers with known auditory problems that prevent participation in MT.

Moreover parents/caregivers with a documented mental illness or cognitive impairment that prevents them from being able to complete the study intervention or outcome assessments.

* Parents/caregivers of premature infants in palliative or end-of-life care, infants with known hearing impairment, or infants in the custody of social services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Postpartum depression | It will be measured during the first week of hospitalization (baseline measurement) and at weeks 1, 2, and 3 of the intervention.
  Postpartum depression will be assessed with the Edinburgh Postnatal Depression Scale (EPDS). This scale has values between 0 to 30 points. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Anxiety | It will be measured during the first week of hospitalization (baseline measurement) and at weeks 2 and 3 of the intervention.
  Anxiety will be assessed with the Generalized Anxiety Disorder Scale (GAD-7). Minimum and maximum possible scores of 0 and 21 respectively. Higher scores mean a worse outcome.
Well-being | It will be measured during the first week of hospitalization (baseline measurement) and at weeks 2 and 3 of the intervention.
  The Warwick Edinburgh Mental Well-Being Scale (WEMWBS) will be employed to assess well-being. Minimum and maximum possible scores of 14 and 70 respectively. Higher scores mean a better wellbeing.
Resilience | It will be measured during the first week of hospitalization (baseline measurement) and at week 3 of the intervention.
  Resilience will be assessed with the Brief Resilience Scale (BRS). Participants respond on a 5-point Likert scale, ranging from 1 (Strongly Disagree) to 5 (Strongly Agree) and giving a range from 6-30. Higher scores mean a better resilience.
Stress | It will be measured during the first week of hospitalization (baseline measurement) and at week 3 of the intervention.
  Stress will be assessed with the 10-item Perceived Stress Scale (PSS-10). Answers are then scored on Likert scale from 0 "Never" to 4 "Very often". Higher scores indicate higher levels of perceived stress.
Coping | It will be measured during the first week of hospitalization (baseline measurement) and at week 3 of the intervention.
  Stress response will be assessed with the Brief COPE Inventory (Brief-COPE). Scores are presented on Likert scale from 1 " I haven't been doing this at all" to 4 "I've been doing this a lot".

CONTACTS AND LOCATIONS:
Locations (5):
- Colombia (4):
  - Clínica Iberoamérica en Colombia, Barranquilla, Atlántico
  - Clinica Pediátrica, Bogotá, Cundinamarca
  - Clínica Universitaria Colombia, Bogotá, Cundinamarca
  - Clínica Keralty Ibagué, Ibagué, Tolima Department
- University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No